CLINICAL TRIAL: NCT02922530
Title: Piloting a Novel, Mobile Cognitive Tracking and Training Tool for Patients With Parkinson's Disease (PD)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator departed for another position.
Sponsor: Posit Science Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSC-1010-16
Record Dates: First submitted 2016-09-29; First posted 2016-10-04 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Experimental Treatment (Experimental): Computerized plasticity-based adaptive cognitive training requiring up to a maximum of 80 treatment sessions, up to 7 sessions per week, 15-60 minutes per session
  Interventions: Other: Computerized Plasticity-based Adaptive Cognitive Training
- Active Comparator (Active Comparator): Commercially available computerized training requiring up to a maximum of 80 treatment sessions, up to 7 sessions per week, 15-60 minutes per session.
  Interventions: Other: Commercially available computerized training

INTERVENTIONS:
Other: Computerized Plasticity-based Adaptive Cognitive Training
  Arms: Experimental Treatment
Other: Commercially available computerized training
  Arms: Active Comparator

SUMMARY:
The overall goal of this research proposal is to develop an adjunct to standard treatments that 'correct' disrupted neural circuitry in Parkinson's Disease (PD) patients. Directly treating these core deficits via targeted behavioral training should slow the progression of PD, assure greater resilience against future decline, and improve the quality of life of many living with PD. The purpose of this exploratory research study is to determine the benefits, if any, of the mobile device-based treatment described above in individuals with PD.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet diagnostic criteria for Parkinson's Disease with mild-to-moderate stage
* Participants must be fluent English speakers
* Participants must have the capability of completing the study as assessed by intact global cognition
* Participants must be able to engage with computerized cognitive tasks as required in the study
* Participants must have normal vision (or corrected to normal vision)
* Participants must have adequate hearing acuity
* Participants must have the motor capacity to use an iPad or mobile device
* Participants must be willing to commit to the time requirements of the study
* Participants must obtain benefit on dopaminergic treatment (dopamine agonist or levodopa) and be on a stable dose for at least one month prior to screening
* Participant must have access to wireless internet connectivity
* Participant must have at least mild depression as assessed by Beck Depression Inventory (BDI-II)

Exclusion Criteria:

* Participants who are unable to perform neuropsychological assessments in the opinion of the evaluating staff person
* Participants who cannot comprehend or follow instructions, in the opinion of the consenting staff person
* Participants who are not capable of giving informed consent, in the opinion of the consenting staff person
* Participants who show signs of intoxication due to current substance abuse (including alcohol and/or illegal drugs) during any in person visit
* Participants with history of significant medical diseases or multiple neurological events of the head
* Participants with serious or unstable medical illness
* Participants with history or current diagnosis of the following Diagnostic and Statistical Manual of Mental Disorders (DSM-5) psychiatric illness: organic mental disorder, schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorder not otherwise specific, bipolar disorder, substance dependence, substance abuse (< 1 year) (subjects with co-occurring post-traumatic stress disorder and related disorders are eligible for participation) as diagnosed through medical history
* Participants with history of seizure disorder
* Participants who are pregnant
* Participants who experience frequent falls (several times a week)
* Participants with severe dyskinesia
* Participants with active suicidal ideations or behaviors as measured by the Columbia-Suicide Severity Rating Scale (C-SSRS)
* Participants enrolled in a concurrent clinical trial involving an investigational pharmaceutical, nutraceutical, medical device, or behavioral treatment that could affect the outcome of this study
* Participant is using computer-based cognitive training programs or has used it within a month of the consent date

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change scores for depressive symptoms using Beck Depression Scale (BDI-II) | At 3 months and 6 months
Change scores for Quality of Life using Parkinson's Disease Questionnaire (PDQ-39) | At 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alit Stark-Inbar, PhD, Principal Investigator — Posit Science Corporation; Mouna Attarha, PhD, Principal Investigator — Posit Science Corporation